CLINICAL TRIAL: NCT04612218
Title: Biomarkers for Initiating Onsite and Faster Ambulance Stroke Therapies (BIO-FAST)
Brief Title: Biomarkers for Initiating Onsite and Faster Ambulance Stroke Therapies
Acronym: BIO-FAST
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Virgen Macarena (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other); Hospital Alta Resolución Sierra Norte (Unknown); Hospital San Juan de Dios Aljarafe (Unknown); Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Joan Montaner Villalonga, Head Department of Neurology, Hospital Universitario Virgen Macarena
Other Study IDs: BIO-FAST
Record Dates: First submitted 2020-10-23; First posted 2020-11-02 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Stroke; Ischemic Stroke; Hemorrhagic Stroke
Keywords: blood biomarkers; stroke diagnosis; stroke; biomarkers; reperfusion therapies; acute stroke therapy; prehospital stroke management
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is the first cause of death among Spanish women and main cause of disability. Reperfusion therapies of the occluded artery remain the only useful approach in acute ischemic stroke. However, the efficacy of these strategies is highly time-dependent and due to the need of neuroimaging (CT or MRI) to differentiate between ischemic and hemorrhagic stroke, impossible to be performed at the pre-hospital level. The investigators aim to set-up a point of-care (POC) device to validate a biomarker panel differentiating ischemic and hemorrhagic stroke at the pre-hospital level using a blood sample and to validate a second biomarker panel for the early identification of patients with large vessel occlusions (LVO), which are candidates for mechanical thrombectomy. For that, the investigators will recruit a 300 patients' cohort with pre-hospital blood samples using available POCs for each of those markers.

ELIGIBILITY:
Inclusion Criteria:

* I.1: Patients > 18 years old.
* I.2: Stroke code activated by the coordinator centre.
* I.3: < 6 hours from symptoms onset. In the case of stroke with uncertain chronology or wake-up stroke, the initial time will be considered as the last moment the patient was seen fine.

Exclusion Criteria:

* E.1: Prehospital diagnosis different of stroke.
* E.2: Impossibility of getting a prehospital blood sample.
* E.3: Refusal to provide the informed consent by the patient/relative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old, in whom health care services activate a stroke code, and the patient is transferred to the reference centre, within 6 hours from symptoms onset.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Stroke subtype diagnostic accuracy | through study completion, an average of 2 years
  Stroke subtype diagnostic (% ischemic versus % hemorrhagic and % stroke mimics) will be determined by clinical and neuroimaging criteria at hospital arrival and compared with diagnostic accuracy of a blood biomarkers based test
Reperfusion rates | through study completion, an average of 2 years
Times to reperfusion | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joan Montaner, PhD, Study Chair — Hospital Universitario Virgen Macarena
Locations (4):
- Spain (4):
  - Hospital de Alta Resolución Sierra Norte, Seville
  - Hospital San Juan de Dios Aljarafe, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville